CLINICAL TRIAL: NCT03258021
Title: The Use of TTFields for Newly Diagnosed GBM Patients in Germany in Routine Clinical Care - TIGER Study
Brief Title: TTFields In GErmany in Routine Clinical Care
Acronym: TIGER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 05.07.2017
Record Dates: First submitted 2017-08-02; First posted 2017-08-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; GBM; Tumor-treating fields; TTFields
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- GBM with indication for TTFields: newly diagnosed GBM with clinical indication for TTFields
  Interventions: Device: TTFields

INTERVENTIONS:
Device: TTFields — Tumor treating fields (TTFields) help slow down or stop glioblastoma cancer cells from dividing by disrupting dividing mechanism of cancer cells leading to apoptosis. TTFields are low-intensity, intermediate frequency, alternating electric fields delivered continuously through adhesive patches, called transducer arrays, to the area of the brain where the GBM tumor is located. These transducer arrays are applied to the scalp and are connected to the wearable and portable device. TTFields are approved for the treatment of newly diagnosed and recurrent GBM.

SUMMARY:
The purpose of this post-authorisation medical device study is to obtain real life data on the use of tumor-treating fields (TTFields) in patients with newly diagnosed GBM in routine clinical care in Germany. Patients with newly diagnosed GBM and clinical indication for TTFields treatment will be enrolled in the study after signing Informed consent to use their data and process it centrally for research purposes. The clinical indication for TTFields is one of the inclusion criteria and is defined prior to inclusion by the treating physician. The patient's decision regarding TTFields treatment is part of the observation and will be assessed within the baseline visit.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common malignant primary tumor of the brain. The current standard of care for patients with newly diagnosed GBM consists of maximal surgical resection, approx. 60 Gy of radiotherapy together with chemotherapy using temozolomide (TMZ), followed by maintenance TMZ for 6 months. This treatment scheme was shown to extend median survival from 12.1 to 14.6 months compared to surgery and radiotherapy alone. This survival was essentially unchanged since 2005 despite numerous clinical Phase 3 trials conducted.

Although immense efforts were made over the years with different treatment strategies, the survival of patients with newly diagnosed GBM remained very poor until recently. Tumor-treating fields (TTFields) are low-intensity, intermediate frequency, alternating electric fields delivered continuously through adhesive patches, called transducer arrays, to the area of the brain where the GBM tumor is located and help slow down or stop glioblastoma cancer cells from dividing. These transducer arrays are applied to the scalp and are connected to the wearable and portable device.

TTFields are the first treatment since 2005 to demonstrate significantly extended median overall survival and significantly improved long-term survival (one to five year survival rates) compared to the current standard of care. In addition, TTFields significantly extended progression-free survival.

In the Phase 3 trial in newly diagnosed GBM (trial EF-14) the results demonstrated that the addition of TTFields to maintenance TMZ significantly extends both, median and long term survival, as well as progression free survival of patients with newly diagnosed GBM. The magnitude of survival benefit seen is even better to that seen for addition of TMZ to radiation, which established TMZ as the standard of care for 1st line GBM treatment in 2005. Quality of life (QoL) was maintained with the use of TTFields + TMZ in patients for whom 12 months of QoL data were available. The addition of TTFields to TMZ therapy in patients with newly diagnosed glioblastoma was not associated with any significant increase in systemic toxic effects compared with TMZ therapy alone. The most commonly reported side effect from the delivery of TTFields was a mild-to-moderate skin irritation beneath the transducer arrays.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed histologically confirmed GBM (WHO-Grade IV)
* Patient within first 3 cycles of first-line tumor-specific maintenance chemotherapy
* ≥ 18 years of age
* Clinical indication for TTFields treatment
* Given informed consent for use and processing of data

Exclusion Criteria:

* Present or planned pregnancy
* Significant additional neurological disease (e.g. significantly increased intracerebral pressure (ICP) with a significant midline shift of the brain)
* Active implanted medical device (e.g. deep brain stimulator)
* Documented allergy to conductive hydrogel
* Skull defect (e.g. missing bone with no replacement, bullet fragments in the skull)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed GBM with clinical indication for TTFields treatment, as indicated by the treating physician, will be included in the study, provided all inclusion and no exclusion criteria are met and written consent is given to use and process their routine clinical data according to data privacy standards.
Sampling Method: Non-Probability Sample
Enrollment: 710 (Actual)
Dates: Start 2017-08-31 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Time to death of any cause (overall survival (OS)) from diagnosis | through study completion, an average of 18 months (mean FU time)
  Time to death of any cause (overall survival (OS)) from diagnosis is measured using the patient data from date of enrollment until the date of death from any cause
Number of TTFields treatment-related serious adverse events (SAEs) standardized to one year of FU time | through study completion, an average of 18 months (mean follow-up time)
  Number of TTFields treatment-related SAEs standardized to one year of follow-up (FU) is measured using the collection of SAEs during the follow-up period
Number of SAEs after start of TTFields treatment | through study completion, an average of 18 months (mean follow-up time)
  Number of SAEs after start of TTFields treatment is measured using the collection of SAEs at the follow-up period
Time of usage (compliance) of TTFields treatment over time | through study completion, an average of 18 months (mean follow-up time)
  Time of usage (compliance) of TTFields treatment over time is measured using the treatment compliance report at the Follow-up period
Time to first progression of GBM (progression-free survival (PFS)), defined within radiological and/or clinical/neurological assessment during routine clinical care in patients who started TTFields treatment at baseline | through study completion, an average of 18 months (mean follow-up time)
  Time to first progression of GBM (progression-free survival (PFS)), defined within radiological and/or clinical/neurological assessment during routine clinical care in patients who started TTFields treatment at baseline from date of enrollment until the date of first progression of GBM
Changes in quality of life at month 2 and month 4 after start of TTFields treatment compared to baseline in patients who started TTFields treatment at baseline | month 2 and month 4 after start of TTFields treatment compared to baseline in patients who started TTFields treatment at baseline
  Changes in quality of life assessed via questionnaires EORTC Quality of life questionnaires (QLQ) QLQ-C30 and BN20 after start of TTFields treatment compared to baseline in patients who started TTFields treatment at baseline is measured using the QoL questionnaires at months two and four after start of TTFields treatment
Patients' reason(s) for refusing TTFields at baseline | baseline
  Patients' reason(s) for refusing TTFields is measured using a study specific questionnaire at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Bähr, Prof., Principal Investigator — Clinical center Aschaffenburg-Alzenau, Aschaffenburg, Germany
Locations (1):
- Clinical center Aschaffenburg-Alzenau, Aschaffenburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolecek TA, Propp JM, Stroup NE, Kruchko C. CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2005-2009. Neuro Oncol. 2012 Nov;14 Suppl 5(Suppl 5):v1-49. doi: 10.1093/neuonc/nos218. No abstract available. PMID 23095881
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Kesari S, Ram Z; EF-14 Trial Investigators. Tumor-treating fields plus chemotherapy versus chemotherapy alone for glioblastoma at first recurrence: a post hoc analysis of the EF-14 trial. CNS Oncol. 2017 Jul;6(3):185-193. doi: 10.2217/cns-2016-0049. Epub 2017 Apr 12. PMID 28399638
- [Background] Stupp R, Wong ET, Kanner AA, Steinberg D, Engelhard H, Heidecke V, Kirson ED, Taillibert S, Liebermann F, Dbaly V, Ram Z, Villano JL, Rainov N, Weinberg U, Schiff D, Kunschner L, Raizer J, Honnorat J, Sloan A, Malkin M, Landolfi JC, Payer F, Mehdorn M, Weil RJ, Pannullo SC, Westphal M, Smrcka M, Chin L, Kostron H, Hofer S, Bruce J, Cosgrove R, Paleologous N, Palti Y, Gutin PH. NovoTTF-100A versus physician's choice chemotherapy in recurrent glioblastoma: a randomised phase III trial of a novel treatment modality. Eur J Cancer. 2012 Sep;48(14):2192-202. doi: 10.1016/j.ejca.2012.04.011. Epub 2012 May 18. PMID 22608262
- [Background] Mrugala MM, Engelhard HH, Dinh Tran D, Kew Y, Cavaliere R, Villano JL, Annenelie Bota D, Rudnick J, Love Sumrall A, Zhu JJ, Butowski N. Clinical practice experience with NovoTTF-100A system for glioblastoma: The Patient Registry Dataset (PRiDe). Semin Oncol. 2014 Oct;41 Suppl 6:S4-S13. doi: 10.1053/j.seminoncol.2014.09.010. Epub 2014 Sep 16. PMID 25213869
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Giladi M, Schneiderman RS, Voloshin T, Porat Y, Munster M, Blat R, Sherbo S, Bomzon Z, Urman N, Itzhaki A, Cahal S, Shteingauz A, Chaudhry A, Kirson ED, Weinberg U, Palti Y. Mitotic Spindle Disruption by Alternating Electric Fields Leads to Improper Chromosome Segregation and Mitotic Catastrophe in Cancer Cells. Sci Rep. 2015 Dec 11;5:18046. doi: 10.1038/srep18046. PMID 26658786
- [Background] Gera N, Yang A, Holtzman TS, Lee SX, Wong ET, Swanson KD. Tumor treating fields perturb the localization of septins and cause aberrant mitotic exit. PLoS One. 2015 May 26;10(5):e0125269. doi: 10.1371/journal.pone.0125269. eCollection 2015. PMID 26010837
- [Background] Kanner AA, Wong ET, Villano JL, Ram Z; EF-11 Investigators. Post Hoc analyses of intention-to-treat population in phase III comparison of NovoTTF-100A system versus best physician's choice chemotherapy. Semin Oncol. 2014 Oct;41 Suppl 6:S25-34. doi: 10.1053/j.seminoncol.2014.09.008. Epub 2014 Sep 16. PMID 25213871
- [Background] Stupp R, Taillibert S, Kanner A, Read W, Steinberg D, Lhermitte B, Toms S, Idbaih A, Ahluwalia MS, Fink K, Di Meco F, Lieberman F, Zhu JJ, Stragliotto G, Tran D, Brem S, Hottinger A, Kirson ED, Lavy-Shahaf G, Weinberg U, Kim CY, Paek SH, Nicholas G, Bruna J, Hirte H, Weller M, Palti Y, Hegi ME, Ram Z. Effect of Tumor-Treating Fields Plus Maintenance Temozolomide vs Maintenance Temozolomide Alone on Survival in Patients With Glioblastoma: A Randomized Clinical Trial. JAMA. 2017 Dec 19;318(23):2306-2316. doi: 10.1001/jama.2017.18718. PMID 29260225